CLINICAL TRIAL: NCT01870609
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of VS-6063 in Subjects With Malignant Pleural Mesothelioma
Brief Title: Placebo Controlled Study of VS-6063 in Subjects With Malignant Pleural Mesothelioma
Acronym: COMMAND
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis-DSMB stated good safety profile but lack of efficacy
Sponsor: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VS-6063-202
Record Dates: First submitted 2013-05-29; First posted 2013-06-06 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-03

CONDITIONS: Malignant Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — defactinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- defactinib (VS-6063) (Active Comparator): 2 x 200 mg defactinib (VS-6063) tablets, administered orally, twice daily
  Interventions: Drug: defactinib (VS-6063)
- Placebo (Placebo Comparator): 2 placebo tablets, administered orally, twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: defactinib (VS-6063)
  Arms: defactinib (VS-6063)
Drug: Placebo — Sugar pill manufactured to mimic defactinib tablet
  Arms: Placebo

SUMMARY:
This study is a Phase 2, randomized, double-blind, placebo-controlled, multicenter study of defactinib (VS-6063) in subjects with malignant pleural mesothelioma (MPM) who have not progressed (confirmed partial response or stable disease) following ≥ 4 cycles of treatment with pemetrexed/cisplatin or pemetrexed/carboplatin. Prior to entry and randomization to the study, each subject must have tumor Merlin status(high or low) established by immunohistochemistry performed at a central laboratory. Subjects will be randomized in a 1:1 ratio to receive oral VS-6063 400 mg twice per day, or matched placebo. Randomization will be stratified by tumor Merlin status (high versus low). Progression will be assessed both locally and by central review using the Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1. Subjects will continue to receive treatment until disease progression or other discontinuation criteria are met. Following documentation of nonfatal disease progression, all subjects will be followed for overall survival by telephone contact every 2 months until end of life or the close of the study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able to understand and give written informed consent and comply with study procedures.
* 2. Histologically proven diagnosis of MPM. All subjects must have biopsy material (archival tissue is acceptable) available for immunohistochemistry determination of Merlin status prior to enrollment.
* 3. Evaluable disease, or measurable disease as assessed by RECIST version 1.1.
* 4. Received only one prior chemotherapy regimen consisting of ≥ 4 cycles of pemetrexed/cisplatin or pemetrexed/carboplatin; subjects must have documentation of an ongoing response (confirmed PR or SD) following completion of this regimen. Subjects changing from cisplatin to carboplatin or vice versa within the same course of treatment because of platinum toxicity will be considered to have had first-line chemotherapy. Note: Subjects may have undergone previous surgical resection of their disease providing it was completed prior to initiation of chemotherapy.
* 5. Received last dose of prior chemotherapy within ≤ 6 weeks of first dose of VS-6063.
* 6. Have completed baseline quality of life evaluation as assessed by LCSS modified for mesothelioma
* 7. Age ≥18 years.
* 8. Life expectancy ≥3 months.
* 9. All prior cytotoxic toxicities must have resolved to grade ≤ 1 prior to randomization.
* 10. Performance status according to the Karnofsky Scale of ≥ 70% (after palliative measures such as pleural drainage).
* 11. Corrected QT interval (QTc) < 470 ms (as calculated by the Fridericia correction formula).
* 12. Adequate bone marrow function (hemoglobin ≥ 9.0 g/dL; platelets ≥ 100 x 109/L; absolute neutrophil count [ANC] ≥ 1.5 x 109/L) without the use of hematopoietic growth factors.
* 13. Adequate renal function (creatinine ≤ 1.5 x ULN [upper limit of normal] or glomerular filtration rate of ≥ 50mL/min).
* 14. Adequate hepatic function (total bilirubin ≤ 1.5 x ULN for the institution; aspartate transaminase [AST] and alanine transaminase [ALT] ≤ 2.5 x ULN).
* 15. Men and women of childbearing potential must agree to use adequate contraception(double barrier birth control) for the duration of study therapy and for 3 months after the last dose of VS-6063.

Exclusion Criteria:

* 1. Currently enrolled in (or completed within 30 days before study drug administration)another investigational drug study.
* 2. GI condition that could interfere with the swallowing or absorption of study drug.
* 3. History of upper GI bleeding, ulceration, or perforation within 12 months prior to the first dose of study drug.
* 4. Known history of Gilbert's Syndrome.
* 5. Known history of stroke or cerebrovascular accident within 6 months prior to the first dose of study drug.
* 6. Subjects with known infection with human immunodeficiency virus or Acquired Immune Deficiency Syndrome (testing not required).
* 7. Subjects with known infection with hepatitis A, B or C (testing not required).
* 8. Any evidence of serious active infections.
* 9. Major surgery within 28 days prior to the first dose of study drug.
* 10. Uncontrolled or severe concurrent medical condition (including uncontrolled brain metastases). Stable brain metastases either previously treated or being treated with a stable dose of steroids and/or anticonvulsants (no dose change within 28 days prior to the first dose of study drug) will be allowed.
* 11. Uncontrolled or severe cardiovascular disease, including myocardial infarct or unstable angina within 6 months prior to study treatment, New York Heart Association Class II or greater congestive heart failure, serious arrhythmias requiring medication for treatment, clinically significant pericardial disease, or cardiac amyloidosis.
* 12 Known history of malignant hypertension.
* 13. Psychiatric illness or social situations that would limit compliance with study requirements.
* 14. History of another invasive malignancy in the last 5 years. Adequately treated noninvasive,non-melanoma skin cancers as well as in situ carcinoma of the cervix within the last 5 years will be allowed.
* 15. Prior treatment with drugs an FAK inhibitor.
* 16. Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2013-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Compare the overall survival (OS) in subjects with malignant pleural mesothelioma receiving defactinib (VS-6063) or placebo | From randomization to end of life, an expected average of 12 months
  The median duration of OS will be estimated based on the 50th percentile of the Kaplan-Meier distribution
Compare the progression free survival (PFS) in subjects with malignant pleural mesothelioma receiving defactinib (VS-6063) or placebo | From date of randomization to earliest documented date of progression, an expected average of 4 months
  PFS will be calculated based on the stratified log-rank test, and will use Kaplan-Meier estimation methods for estimation of summary statistics

SECONDARY OUTCOMES:
To assess Quality of Life (QoL) in subjects treated with defactinib (VS-6063) or placebo using the Lung Cancer Symptom Scale modified for mesothelioma (LCSS-Meso) | Every 3-4 weeks from baseline through end of treatment, an expected average of 4 months
  QoL will be assessed using the LCSS-Meso. The LCSS-Meso total score will be analyzed through a comparison of median area under the curve (AUC) between the 2 treatment groups using a Wilcoxon test.
To determine the objective response rate (ORR) in subjects receiving defactinib (VS-6063) or placebo. | Every 6-8 weeks from baseline through end of treatment, an expected average of 4 months
  ORR is measured as the best overall response assessed by central review using Response Evaluation Criteria In Solid Tumors (RECIST), version 1.1.

OTHER OUTCOMES:
Determine the time to new lesion in subjects receiving defactinib (VS-6063) or placebo | Every 6-8 weeks from baseline until end of treatment, an expected average of 4 months
  Time to new lesion will be calculated from the date of randomization to the time of CT scan documenting a new lesion or date of other unambiguous indicator of new lesion development.
Evaluate the relationship of defactinib (VS-6063) pharmacokinetics (PK) and outcome | Time points at Week 4, Week 7, Week 10 and Week 13
  PK parameters, including but not limited to plasma concentration, AUC (Area Under Curve) 0-t, Cmax, Tmax, and T1/2, compared with outcome
Evaluate the population pharmacokinetics of defactinib (VS-6063) in subjects with malignant pleural mesothelioma | Time points at Week 4, Week 7, Week 10 and Week 13
  PK parameters, including but not limited to plasma concentration, AUC (Area Under Curve) 0-t, Cmax, Tmax, and T1/2
Evaluate the safety and tolerability of defactinib (VS-6063) in subjects with malignant pleural mesothelioma | From start of treatment to end of treatment, an expected average of 4 months
  Adverse events and their frequency, duration and severity, physical examination, laboratory parameters, vital signs and ECG change monitoring as determined based on CTCAE (Common Toxicity Criteria for Adverse Effects) 4.03
To collect EuroQol 5-Dimensional Health Questionnaire (EQ-5D) for health economics purposes | Every 3-4 weeks from baseline through end of treatment, an expected average of 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, Study Chair — Verastem, Inc.
Locations (73):
- United States (12):
  - University of California San Francisco Medical Center, San Francisco, California
  - Cleveland Clinic Florida, Weston, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Abramson Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
- Australia (8):
  - Peninsula Oncology Centre, Frankston, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
  - Chris O'Brien Lifehouse at RPA, Camperdown
  - Monash Cancer Center, East Bentlrigh
  - Epworth Hospital, Melbourne
  - Northern Cancer Institute, Sydney
  - Calvary Mater Newcastle, Waratah
  - Princess Alexandra Hospital +61(0)7 3176 5054, Woolloongabba
- Belgium (5):
  - UCL - St. Luc, Brussels
  - Antwerp University Hospital, Edegem
  - University Hopsital Ghent, Ghent
  - Universitaire Ziekenhuizen Leuven (University Hospitals Leuven), Leuven
  - CHU Liege - Sart Tilman, Liège
- Princess Margaret Hospital, Toronto, Ontario, Canada
- France (3):
  - CHRU, Lille, Lille
  - Hôpitaux de Marseille, Marseille
  - Gustave Roussy, Villejuif
- Italy (2):
  - Cliniche Humanitas Gavazzeni, Bergamo
  - Istituto Oncologico Veneto, Padua
- Japan (6):
  - Kyushu Cancer Center, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Hyogo College of Medicine, Hyōgo
  - Okayama Rousai Hospital, Okayama
  - Kinki University Hospital, Osaka
  - Juntendo University, Tokyo
- Netherlands (4):
  - Stichting Het Nederlands Kanker Instituut-Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Medisch Spectrum Twente, Enschede, Enschede
  - Atrium MC, Heerlen
  - Erasmus MC, Rotterdam
- New Zealand (2):
  - Auckland Oncology Research Centre, Auckland
  - Canterbury Regional Cancer & Haematology Service, Christchurch
- Norwegian Radium Hospital, Oslo, Norway
- Centrum Pulmonologii Ii Torakochirurgii w Bystrej, Bystra, Poland
- South Africa (3):
  - Iatros International / Bloemfontein Medi-Clinic, Bloemfontein, Free State
  - The Medical Oncology Centre of Rosebank, Johannesburg
  - Mary Potter Oncology Center, Little Company of Mary Hospital, Pretoria
- Spain (4):
  - Institut Oncològic del Vallés Consorci Hospitalari Parc Tauli, Barcelona
  - Vall d'Hebron University Hospital, Barcelona
  - Ensayos Clínicos Oncología, Madrid
  - Hospital Madrid Norte- Sanchinarro, Centro Integral Oncológico Clara Campal (CIOCC), Madrid
- Sweden (3):
  - Skane University Hospital, Lund
  - Karolinska University Hospital, Stockholm
  - University Hospital, Uppsala
- United Kingdom (18):
  - Clatterbridge Cancer Centre, Bebington, Wirral
  - Southmead Hospital, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Velindre Hospital Cardiff, Cardiff
  - Broomfield Hospital, Chelmsford
  - Tayside Cancer Centre, Dundee
  - Beatson Oncology Centre, Glasgow
  - Royal Surrey County Hospital, Guildford
  - Castle Hill Hospital, Hull
  - Kent Oncology Centre, Maidstone Hospital, Kent
  - University of Leicester, Leicester
  - Guys Hospital, London
  - St. Bartholomew's Hospital, London
  - Wythenshawe Hospital, Manchester
  - Freeman Hospital, Newcastle
  - Derriford Hospital, Plymouth
  - Weston Park Hospital, Sheffield
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Fennell DA, Baas P, Taylor P, Nowak AK, Gilligan D, Nakano T, Pachter JA, Weaver DT, Scherpereel A, Pavlakis N, van Meerbeeck JP, Cedres S, Nolan L, Kindler H, Aerts JGJV. Maintenance Defactinib Versus Placebo After First-Line Chemotherapy in Patients With Merlin-Stratified Pleural Mesothelioma: COMMAND-A Double-Blind, Randomized, Phase II Study. J Clin Oncol. 2019 Apr 1;37(10):790-798. doi: 10.1200/JCO.2018.79.0543. Epub 2019 Feb 20. PMID 30785827